CLINICAL TRIAL: NCT02209766
Title: A Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics in Healthy Male Japanese (Single-blind, Randomized, Placebo-controlled) and Caucasian (Open-label) Subjects After Single and Once Daily Multiple Oral Doses of D5884
Brief Title: A Ph1 Study in Healthy Male Japanese and Caucasian After Single and Multiple Doses of D5884(Omega-3-carboxylic Acids)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D5881C00005
Record Dates: First submitted 2014-08-01; First posted 2014-08-06 (Estimated); Results first posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; D5884; Japanese; Caucasian

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- D5884 (Experimental): D5884 capsule, Per oral(po)
  Interventions: Drug: D5884
- Placebo (Placebo Comparator): Placebo capsule, po
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D5884 — 1st cohort: Dose 1(2g) D5884(n=6) in Japanese 2nd cohort: Dose 2(4g) D5884(n=6) in Japanese 3rd cohort: Dose 2(4g) D5884(n=6) in Caucasian
  Arms: D5884
Drug: Placebo — 1. st cohort: Dose 1(2g) D5884(n=3) in Japanese
  2. nd cohort: Dose 2(4g) D5884(n=3) in Japanese
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety, tolerability and pharmacokinetics of D5884 following administration of single and multiple doses in healthy male Japanese subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single-centre study that plans to enrol 3 cohorts in 3 study arms (Study Arms A, B and C). Study Arms A and B will be comprised of cohorts of healthy male Japanese subjects in randomised, single-blind, placebo-controlled, single and multiple dose parallel studies and Study Arm C will be comprised of a cohort of healthy male Caucasian subjects in a single and multiple dose open-label study.

Two dose levels, 2 and 4 g D5884, will be investigated in healthy male Japanese subjects. Up to 18 healthy male Japanese subjects aged 20 to 45 years, inclusive, will be enrolled in 2 cohorts (Study Arms A and B) and up to 6 healthy male Caucasian subjects will be enrolled in a 3rd cohort (Study Arm C). Each subject will participate in 1 cohort only.

Following a screening period of a maximum of 42 days, subjects will reside at the study facility for 18 nights starting from the day before dosing (Day -1) to Day 18 (day of discharge). The follow-up period after dosing will be 8 (±2) days after last dose. Dose administration in all 3 study arms will be done in the following sequence: a single dose of D5884 or placebo will be administered; this will be followed by a 2-day washout period; after the washout period, multiple doses of D5884 or placebo will be administered, once daily for 14 consecutive days. The 1st cohort (Study Arm A) will receive 2 g D5884 (n=6) or placebo (n=3), the 2nd cohort (Study Arm B) will receive 4 g D5884 (n=6) or placebo (n=3) and the 3rd cohort (Study Arm C) will receive 4 g D5884 (n=6).

The PK analysis included all evaluable PK data appropriate for the evaluation of interest (eg, with no major protocol deviations or violations thought to significantly affect the PK of the drug) from all subjects who received D5884.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male, 20 to 45 years of age (inclusive)
2. Body mass index (BMI) ≥18.5 and ≤25 kg/m2 for Japanese subjects, ≥18.5 and ≤30 kg/m2 for Caucasian subjects. BMI calculations to be conducted on height and weight values obtained at Visit 1
3. Medically healthy with clinically insignificant screening results (eg, laboratory profile, medical history, ECGs, physical examination). Haemoglobin has to be ≥ the lower limit of the study site reference range, 12-lead ECG must have QT interval corrected for heart rate using Fridericia's formula(QTcF) >340 msec and <450 msec
4. No habitual use of drug(s) and non-tobacco/nicotine-containing products for a minimum of 6 months prior to dosing
5. Subjects must be willing and able to give written informed consent by signing an Institutional Review Board(IRB)-approved informed consent form (ICF) prior to admission to this study and follow the restrictions and procedures outlined for the study.
6. Mean fasting Triglyceride(TG) at -4 and -2 weeks of <150 mg/dL, and %TG change of <30% between Weeks -4 and -2

Exclusion Criteria:

1. Participation in another clinical study with an investigational product(IP) during the 4 months prior to enrolment
2. Past history of psychological or physical disorder which may affect the objectives of this study, in the opinion of the PI
3. An individual who has abnormal laboratory values (ie, suggesting hepatic, renal, cardiovascular or endocrine disorders or diabetes mellitus), or an inappropriate current or past medical history for participation based on the decision of the principal investigator(PI)
4. A history or presence of significant cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease
5. A positive urine drug/alcohol test at screening or admission (Visit 3, Day -1). (The drug test includes testing for phencyclidine, benzodiazepine, cocaine, amphetamines, cannabis, opiates, barbiturates and tricyclic anti-depressants. The alcohol test is an alcohol breath assessment.)
6. A positive test for syphilis, human immunodeficiency virus, hepatitis B surface antigen or hepatitis C virus antibodies.
7. Had used fish oil, other EPA- and/or DHA-containing supplements within 2 months of the planned time of admission
8. Current evidence, or a history of alcoholism or drug abuse within the 2 years prior to admission
9. A known sensitivity or allergy to soybeans, fish and/or shellfish
10. A hypersensitivity or idiosyncratic reaction to compounds related to EPA and/or DHA
11. Had used any prescription medication within 14 days prior to admission
12. Had used any over-the-counter (OTC) medication, including herbal products (bromelains, danshen, dong quai [Angelica sinensis], garlic, ginko biloba, ginseng, and St. John's wort), within the 7 days prior to admission
13. Had used any drugs known to significantly inhibit [strong or moderate] or induce liver enzymes involved in drug metabolism [cytochrome P450]) within 30 days prior to admission
14. Had donated blood or had had significant blood loss in excess of 200 mL within 1 month prior to admission or in excess of 400 mL within 3 months prior to admission
15. Had donated plasma within 7 days prior to admission
16. History of drug abuse or past history of alcohol abuse or habit of taking nicotine-containing product(s) on a daily basis
17. Those who have difficulty in giving blood during blood sampling via the peripheral vein
18. Any potential subjects who are considered as not eligible for the study in the opinion of the PI and/or the sub-investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Fukase, MD, Principal Investigator — CPC Clinical Trial Hospital
Locations (1):
- CPC Clinical Trial Hospital, Kagoshima, Kagoshima-ken, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 86 male subjects were screened.
Pre-assignment Details: Of the 86 subjects, 43 did not meet the inclusion/exclusion criteria, 14 decided not to participate in the study and 5 had other reasons for declining participation in the study.
Groups:
- 2 g D5884 Japanese; 2 g D5884 Japanese Placebo; 4 g D5884 Japanese; 4g D5844 Japanese Placebo; 4g D5884 Caucasian: Single dose followed by once daily for 14 consecutive days
Period: Overall Study
Arm/Group | 2 g D5884 Japanese | 2 g D5884 Japanese Placebo | 4 g D5884 Japanese | 4g D5844 Japanese Placebo | 4g D5884 Caucasian
Started | 6 | 3 | 6 | 3 | 6
Completed | 6 | 3 | 6 | 2 | 6
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- 4 g D5884 Caucasian; Placebo Japanese: Single dose followed by once daily for 14 consecutive days
- Total: Total of all reporting groups
Arm/Group | 2 g D5884 Japanese | 4 g D5884 Japanese | 4 g D5884 Caucasian | Placebo Japanese | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (8.71) | 28.3 (6.15) | 34.0 (5.25) | 32.3 (6.12) | 30.3 (6.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 6 | 6 | 0 | 6 | 18
  Caucasian | 0 | 0 | 6 | 0 | 6
Weight [Mean (Standard Deviation); unit: kg] | 60.42 (8.109) | 69.08 (7.059) | 72.92 (10.169) | 62.63 (6.371) | 66.26 (9.078)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.67 (0.852) | 22.67 (1.517) | 22.55 (1.724) | 21.40 (1.370) | 21.82 (1.559)

OUTCOME MEASURES:

1. Secondary Outcome: Cmax in Plasma Baseline-adjusted Total Eicosapentaenoic Acid (EPA), Single Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- 2g D5884 Japanese; 4g D5884 Japanese; 4g D5885 Caucasian: Single dose followed by once daily for 14 consecutive days
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 82.22 (45.10) | 220.0 (17.70) | 158.1 (34.98)

2. Secondary Outcome: Tmax in Plasma Baseline-adjusted Total EPA, Single Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Median (Full Range); unit: h
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
h | 5.50 [5.00 to 6.00] | 5.00 [5.00 to 6.00] | 6.00 [5.00 to 8.00]

3. Secondary Outcome: Cmax in Plasma Baseline-adjusted Total Docosahexaenoic Acid (DHA), Single Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 32.04 (69.51) | 90.10 (21.50) | 63.63 (46.12)

4. Secondary Outcome: Tmax in Plasma Baseline-adjusted Total DHA, Single Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Median (Full Range); unit: h
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
h | 5.00 [4.00 to 6.00] | 5.00 [5.00 to 6.00] | 5.00 [5.00 to 6.00]

5. Secondary Outcome: Cmax in Plasma Baseline-adjusted Total EPA, Multiple Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 157.4 (32.73) | 314.8 (26.09) | 238.8 (33.21)

6. Secondary Outcome: Tmax in Plasma Baseline-adjusted Total EPA, Multiple Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Median (Full Range); unit: h
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
h | 5.00 [5.00 to 6.00] | 5.50 [5.00 to 6.00] | 5.00 [5.00 to 7.00]

7. Secondary Outcome: Cmax in Plasma Baseline-adjusted Total DHA, Multiple Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 58.47 (49.15) | 88.21 (89.54) | 101.1 (34.06)

8. Secondary Outcome: Tmax in Plasma Baseline-adjusted Total DHA, Multiple Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Median (Full Range); unit: h
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
h | 5.00 [5.00 to 6.00] | 6.00 [5.00 to 6.00] | 5.00 [5.00 to 6.00]

9. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events (TEAEs), by Treatment (Safety Analysis Set)
Description: Number of patients with treatment-emergent adverse events (TEAEs), by treatment (Safety Analysis Set)
Time Frame: from first dosing (Day1) until follow-up (Day25)
Measure: Number; unit: subjects
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian | Placebo Japanese
Number analyzed (Participants) | 6 | 6 | 6 | 6
subjects
  TEAEs | 2 | 2 | 5 | 2
  TEAEs leading to discontinued | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0

10. Secondary Outcome: AUC(0-tau) in Plasma Baseline-adjusted Total DHA, Multiple Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg*h/mL | 531.2 (75.81) | 621.9 (278.9) | 1044 (48.00)

11. Secondary Outcome: AUC(0-tau) in Plasma Baseline-adjusted Total EPA, Multiple Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg*h/mL | 2072 (39.29) | 4067 (43.52) | 3136 (28.93)

12. Secondary Outcome: AUC(0-tau) in Plasma Baseline-adjusted Total Docosahexaenoic Acid (DHA), Single Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg*h/mL | 138.2 (80.07) | 432.9 (39.97) | 783.2 (78.67)

13. Secondary Outcome: AUC(0-tau) in Plasma Baseline-adjusted Total Eicosapentaenoic Acid (EPA), Single Dose
Time Frame: Day1-3, 4, 7, 11, 14, 17-18 and 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 2g D5884 Japanese | 4g D5884 Japanese | 4g D5885 Caucasian
Number analyzed (Participants) | 6 | 6 | 6
μg*h/mL | 1108 (38.37) | 2213 (31.67) | 2105 (25.70)

ADVERSE EVENTS:
Time Frame: AEs will be collected from randomisation, throughout the treatment period and including the follow-up period. SAEs will be recorded from the time of informed consent.
Arm/Group | 2 g D4884 Japanese | 4 g D4884 Japanese | 4 g D4884 Caucasian | Placebo Japanese
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 5/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 0.166% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 g D4884 Japanese (N=6) | 4 g D4884 Japanese (N=6) | 4 g D4884 Caucasian (N=6) | Placebo Japanese (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALT increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
AST increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less